CLINICAL TRIAL: NCT04732026
Title: PREPARE Work Package 3 -Development of a Serocorrelate of Protection Against GBS - Protocol Harmonisation.
Brief Title: Serocorrelate of Protection Against GBS (PREPARE WP3)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: MU-JHU CARE (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other); University of Liverpool (Other); Assistance Publique - Hôpitaux de Paris (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0021
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Group B Streptococcus Carrier in Childbirth; Group B Streptococcal Infection, Late-Onset; Group B Streptococcal Infection, Early-Onset; Group B Streptococcus Neonatal Sepsis; Group B Strep Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood - target volume 5mls, minimum 1.5mls Maternal serum- target volume 5mls, minimum 1.5mls Infant serum - target volume 2mls, minimum based on infant birthweight Bacterial Isolates - GBS isolates from blood or CSF of infants with invasive GBS disease
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 150 infants with invasive serotype III GBS disease (isolation of GBS from a normally sterile site, i.e. blood or CSF) in the first 90 days of life from six countries (Malawi, Uganda, UK, the Netherlands, Italy and France).
- Controls: 450 infants exposed to serotype III GBS at birth - but who do not develop invasive GBS disease in the first 90 days of life from six countries (Malawi, Uganda, UK, the Netherlands, Italy and France).

SUMMARY:
A multicentre, international case-control study to develop a biobank of sera from 150 cases of serotype III GBS disease and associated clinical information from seven countries (Malawi, Uganda, UK, the Netherlands, Italy and France), with 3:1 (450) serotype matched healthy controls.

DETAILED DESCRIPTION:
Group B Streptococcus (GBS) causes severe infections in young infants across the world. In 2015 it was estimated that there were at least 319,000 infants under three months of age with GBS disease worldwide, resulting in 90,000 deaths and at least 10,000 children with long term disabilities. Around 20% of all pregnant women carry GBS in their vagina and bowel, and babies are exposed to GBS bacteria around the time of birth. The options for prevention are currently limited to offering antibiotics during labour.

A vaccine that could be given to pregnant women has the greatest potential to benefit mothers and babies worldwide. There are vaccines currently being tested in clinical trials, including in pregnant women. Given the complexity, size and costs associated with a phase III trial, it is generally agreed that indirect evidence (correlates) of protection (CoP), based on immunologic data from vaccine and seroepidemiological studies, opsonophagocytic assays and supported by animal models, could be pivotal for vaccine licensure, with effectiveness subsequently confirmed in post-licensure evaluations.

This study aims to develop a biobank of sera from 150 cases of serotype III GBS disease and associated clinical information from seven countries (Malawi, Uganda, UK, the Netherlands, Italy and France) with 3:1 (450) serotype matched healthy controls.

GBS cases will be identified through active surveillance of GBS disease in infants, as part of ongoing epidemiological studies in Uganda, the UK, Italy, France, the Netherlands and Malawi. Upon identification of cases, consent will be requested to obtain a serum sample (1-2 mL of blood collected from infant), the GBS isolate and to collect brief clinical and demographic details. Each site will aim to collect around 50 cases of invasive GBS disease cases (with all samples) over the course of 2 years.

Each site will also recruit approximately 1000 women to have a rectovaginal swab at 35-37 weeks gestation and cord and maternal blood samples at delivery. These women and their infants will be followed up to 90 days of age and considered appropriate controls if the infants are exposed to the same serotype/strain of GBS at delivery as the case - but do not develop GBS the first 90 days of life. We will select 3 controls for every case.

The biorepository will be established at the St George's University of London for all samples from the European Union and Malawi and the MRC/UVRI & LSHTM Uganda Research Unit for Ugandan samples.

ELIGIBILITY:
Inclusion Criteria:

Cases:

Infant 0-90 days of life with GBS identified from a normally sterile site.

Controls:

Healthy infant born to a GBS colonised woman that does not develop GBS disease between birth and 90 days of life.

Exclusion Criteria An infant is not eligible unless a parent/person with parental responsibility gives informed consent.

Max Age: 90 Days | Sex: All
Age Groups: Child
Study Population: The study will enroll infant subjects from the general population who are delivered at one of the six hospital sites.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
To establish a biobank of at least 150 GBS serotype III cases including both the isolate and associated maternal and infant serum. | Over the course of 2 years
  Biobank at St George's, University of London

SECONDARY OUTCOMES:
To determine the quantity of antibody associated with protection against GBS disease | Over the course of 2 years
  Geometric mean and median antibody titres will be calculated for cases and controls and comparisons made as appropriate
To determine the functional antibody associated with protection against GBS disease. | Over the course of 2 years
  Samples will be tested using opsonophagocytosis killing assay for both anti-capsular and anti-protein antibodies.
To demonstrate the relationship between antibody quantity and function in protection against GBS disease | Over the course of 2 years
  To directly compare total antibody concentration titers (measured by multiplex LUMINEX) with opsonophagocytosis from functional antibodies at the time of birth and at the time of disease.
To refine estimates for serocorrelates of protection against GBS disease. | Over the course of 2 years
  To provide initial data on the relationship between antibody and invasive GBS disease risk by estimating the odds ratio of invasive GBS disease for antibody concentrations above various thresholds for STIII
To provide training to participating African laboratories to assure the quality of sample collection and data curation. | Over the course of 2 years
  A South-South partnership between Makerere University John Hopkins Research Collaboration (MUJHU),and Malawi-Liverpool-Wellcome Trust Clinical Research Programme (MLW) to optimise the capacity for conducting clinical trials for maternal immunisation in Sub-Saharan Africa

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, Prof, Principal Investigator — St George's, University of London; Stephen Cose, Dr, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (6):
- Assistance Publique Hopitaux de Paris (AP-HP), Paris, France
- Azienda Ospedaliero-Universitaria di Modena (AOU), Modena, Italy
- Queen Elizabeth Central Hospital College of Medicine, P.O. Box 30096 Chichiri,, Blantyre, Malawi
- Academisch Medisch Centrum,Universiteit van Amsterdam, Amsterdam, Netherlands
- MUJHU - Makerere University Johns Hopkins University Research Collaboration/MUJHU Care Ltd, Kampala, Uganda
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No